CLINICAL TRIAL: NCT03581955
Title: Identification of New Biomarkers of Banana and Tomato Intake
Acronym: BioBanaTom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudine MANACH (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor-Investigator, Claudine MANACH, Principal Investigator, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Organization: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016-A00153-48
Record Dates: First submitted 2017-08-31; First posted 2018-07-10 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Biomarkers; Food Intake
Keywords: biomarkers; diet; banana; tomato; urine; plasma; intake; exposure; metabolomics
MeSH Terms: interventions — Fresubin

STUDY DESIGN:
Intervention Model Description: The present project is a randomized, controlled, crossover study with 12 subjects. A cross-over design has been selected as each subject can serve as his/her own control thereby minimizing variations. The intervention order was randomized. The study design does not allow blinding as intervention is the ingestion of different foods.In this study, we assessed the metabolomic profiles of human biofluids after consumption of two different foods: banana (240g peeled fruit) and tomato (300g fresh fruit) in order to identify novel biomarkers for each food. As a control diet, a high energy high protein drink, Fresubin ® 2kcal fiber (Fresinius kabi) was used. The study comprised three dietary interventions of 4 days each and a wash-out period no shorter than 3 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Banana Cavendish (Experimental): 240g of fruit plus 150ml of Fresubin ® 2kcal fiber neutral flavor
  Interventions: Other: Banana Cavendish
- Control drink (Experimental): 250ml of Fresubin ® 2kcal fiber neutral flavor
  Interventions: Other: Fresubin ® 2kcal fiber neutral flavor
- Tomato (Experimental): 300g of tomato plus of Fresubin ® 2kcal fiber neutral flavor plus 12g of refined sunflower oil.
  Interventions: Other: Tomato

INTERVENTIONS:
Other: Banana Cavendish — 240g of fruit plus 150ml of control drink (Fresubin ® 2kcal fiber neutral flavor)
  Other Names: Test Food
  Arms: Banana Cavendish
Other: Tomato — 300g of raw tomato ("coeur de boeuf") with refined sunflower oil (12g) and 150ml of control drink (Fresubin ® 2kcal fiber neutral flavor).
  Other Names: Test Food
  Arms: Tomato
Other: Fresubin ® 2kcal fiber neutral flavor — 250 ml Fresubin ® 2kcal fiber neutral flavor
  Other Names: Control
  Arms: Control drink

SUMMARY:
The intake of fruits and vegetables has been associated to a lower risk of developing metabolic diseases and cancer. The intake of tomato has been proposed to decrease the risk of prostate cancer while the high content of pro-vitamine A carotenes in banana have shown to alleviate Vitamin A deficiency in different countries. Interestingly in spite of their popularity, there are no biomarkers of banana intake reported in the literature while lycopene is the most frequently used metabolite to indicate tomato consumption however, its limited specificity and between-subjects variation sets doubt of its accuracy. Therefore, the identification of novel biomarkers for both banana and tomato is of great value. Untargeted metabolomics, allows a holistic analysis of the food metabolome allowing a deeper inquiry in the metabolism of different compounds and the recognition of patterns and individual differences that may lead to new hypothesis and further research. Therefore, the aim of the present study is to identify biomarkers of acute intake of banana and tomato using an untargeted approach on urine serum of 12 volunteers that participated in a crossover, randomized, controlled study. Volunteers consumed three different test foods: 1) 240g of banana, 2) 300g of tomato and 3) Fresubin 2kcal as control. Serum and urine samples were collected in kinetics over 24h and processed to be analyzed using LC-QTof analysis. The metabolomics profiles are compared using univariate (ANOVA) and multivariate statistical methods (PCA, PLSDA). The identification of discriminant compounds was performed by tandem mass fragmentation with a high-resolution LTQ-Orbitrab Mass spectrometer and by an extensive inquiry of different online databases.

DETAILED DESCRIPTION:
The rise of metabolomics along with different platforms such as liquid chromatography mass spectrometers (LC-MS) have allowed the assessment of thousands of metabolites simultaneously in biological samples and the recognition of patterns that may constitute a fingerprint of the intake of different foods. Recent studies demonstrated the great potential of metabolomics to discover new biomarkers of intake in intervention and cohort studies.The diversity of compounds found in food metabolomics represents a major challenge and so in an international effort to improve dietary biomarkers identification and validation, the Food Biomarkers Alliance (FOODBALL) has been created. In this project, 22 institutions from 11 different countries will collaborate in three main tasks: 1) Discovery of new dietary biomarker using a metabolomic approach, 2) systemic validation of existing and newly discovered biomarker to achieve a good coverage of food intake in different European populations and 3) exploring biological effects using biomarkers of intake (http://foodmetabolome.org/). With the latter, the necessity of building a chemical library that allows the use of standards for further identification arises. Along with FOODBALL, The Food Compound Exchange (FoodComEx) aims to improve the availability of analytical standards of biological compounds to achieve a better and easier biomarker identification (http://foodcomex.org/).

As part of INRA collaboration to FOODBALL and FoodComEx, the present project attempts to identify biomarkers of banana and tomato intake, through the exploration of the serum and urine metabolome of 12 subjects who consumed these foods following a randomized, controlled, crossover design. The present study was comprised of 3 different intervention periods and a minimum of 3 days washout between interventions. The intervention periods were comprised of 2 run in days, 1 intervention day and 1 post intervention day. In the first day of the run in period, subjects were instructed to avoid the intake of banana or tomato or any of their products; the day prior to the intervention volunteers were asked to avoid the intake of phytochemical rich foods and beverages such as wine, coffee, chocolate, tea, and other plant based foods including banana and tomato.In the morning of the intervention, day subjects arrived in fasting state to the research center at 7.30 am. Volunteers were randomly assigned to one of the three interventions, Fresubin ® 2kcal fiber, 240g of banana plus control drink, or 300g of tomato plus control drink plus 12g of refined sunflower oil. Throughout the intervention, subjects had free access to water, maximum 250ml of water per hour until 6 hours after the intake of the test food.

A trained phlebotomist placed a catheter on the subject's arm before the intake of the test foods to collect the baseline sample. Then four other samples were collected postprandially after 1h, 2h, 4h, and 6h. A total of 7 urine samples were collected. The first void of urine was collected by the subjects at home upon the morning of Day 3 and the rest of the samples after the intake of the test foods as follows: 0-1h, 1h-2h, 2h-4h, 4h-6h. The urine samples corresponding to 6h-12h and 12-24h interval were collected by volunteers at home until the morning after the intake of the food.

After the 6h collection of blood, the peripheral catheter was removed and subjects had lunch composed of white bread and cooked pasta, then subjects were allowed to go home. Before leaving the Investigation center, participants were instructed to prepare a standardized dinner based on pan fried chicken with butter and boiled rice with salt. Volunteers were not allowed to eat or drink anything except water and the standardized dinner.

On the morning of the post intervention day, subjects arrived in fasting state to the research center to give the 24h blood sample and deliver the 06-12h and 12-24h urine collection. Afterward, subjects were served breakfast at the research center and resumed their normal diet until the next run in days of the next intervention period.

Urine samples and serum samples were aliquoted and stored at -80° C until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged 18- 40 years
* BMI >18.5 and < 30 kg/m2
* Willing/able to consume all test foods (tomato, banana, Fresubin drink) and the standardized meals (rice and chicken)

Exclusion Criteria:

* Smokers
* Diagnosed health condition (chronic or infectious disease)
* Taking nutritional supplements (e.g. vitamins, minerals) several times a week.
* Taking medication (oral contraceptive pill is allowed).
* Pregnant, lactating.
* Antibiotics treatment within 3 months prior to intervention.
* Vegetarians, as standardized meals will contain meat.
* Not willing to follow nutritional restrictions, including drinking alcohol during study days
* Not willing/able to give informed consent or to sign informed consent.
* Not affiliated to National Health Insurance.
* Being in exclusion on the National Volunteers Data file or refusing to be registered on the National Volunteers Data file.
* Currently participating or who having got 4500€ in this year to have participated in another clinical trial.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03-26 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-06-16 (Actual)

PRIMARY OUTCOMES:
Changes in metabolite profiles present in blood serum and urine before the dietary intervention (t=0) and in kinetics over 24 hours. | 0-24 hours
  Metabolite profiles analyzed using a non-targeted metabolomics approach with a UPLC-MS platform. Blood serum samples collected at time 0, 1 hour, 2 hours, 4 hours, 6 hours and 24 hours. Urine fractions collected at 0-1 hours, 1-2 hours, 2-4 hours, 4-6 hours, 6-12 hours, 12-24 hours. Identification of biomarkers of acute intake of the foods of interest through the comparison of metabolomes after either single dose of tomato, banana or control drink.

SECONDARY OUTCOMES:
Collection of pools of urine and serum samples after acute intake of tomato or banana to be used as analytical standards or for the identification of specific metabolites of banana or tomato components. | 0-24 hours
  The collection of pools of biofluids that result from this study may be shared with the scientific community through the FoodComEx library in order to be used as an analytical standard or for the identification of metabolites that are specific of banana or tomato intake.

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Manach, Researcher, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- INRA, Clermont-Ferrand, Rhône-Alpes-Auvergne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen MB, Kristensen M, Manach C, Pujos-Guillot E, Poulsen SK, Larsen TM, Astrup A, Dragsted L. Discovery and validation of urinary exposure markers for different plant foods by untargeted metabolomics. Anal Bioanal Chem. 2014 Mar;406(7):1829-44. doi: 10.1007/s00216-013-7498-5. Epub 2014 Jan 4. PMID 24390407
- [Background] Manach C, Hubert J, Llorach R, Scalbert A. The complex links between dietary phytochemicals and human health deciphered by metabolomics. Mol Nutr Food Res. 2009 Oct;53(10):1303-15. doi: 10.1002/mnfr.200800516. PMID 19764066
- [Background] Scalbert A, Brennan L, Manach C, Andres-Lacueva C, Dragsted LO, Draper J, Rappaport SM, van der Hooft JJ, Wishart DS. The food metabolome: a window over dietary exposure. Am J Clin Nutr. 2014 Jun;99(6):1286-308. doi: 10.3945/ajcn.113.076133. Epub 2014 Apr 23. PMID 24760973
- [Background] Re R, Bramley PM, Rice-Evans C. Effects of food processing on flavonoids and lycopene status in a Mediterranean tomato variety. Free Radic Res. 2002 Jul;36(7):803-10. doi: 10.1080/10715760290032584. PMID 12180131
- [Background] Giovannucci E. Tomatoes, tomato-based products, lycopene, and cancer: review of the epidemiologic literature. J Natl Cancer Inst. 1999 Feb 17;91(4):317-31. doi: 10.1093/jnci/91.4.317. PMID 10050865
- [Background] Pereira A, Maraschin M. Banana (Musa spp) from peel to pulp: ethnopharmacology, source of bioactive compounds and its relevance for human health. J Ethnopharmacol. 2015 Feb 3;160:149-63. doi: 10.1016/j.jep.2014.11.008. Epub 2014 Nov 13. PMID 25449450
- [Background] Pujos-Guillot E, Hubert J, Martin JF, Lyan B, Quintana M, Claude S, Chabanas B, Rothwell JA, Bennetau-Pelissero C, Scalbert A, Comte B, Hercberg S, Morand C, Galan P, Manach C. Mass spectrometry-based metabolomics for the discovery of biomarkers of fruit and vegetable intake: citrus fruit as a case study. J Proteome Res. 2013 Apr 5;12(4):1645-59. doi: 10.1021/pr300997c. Epub 2013 Mar 5. PMID 23425595
- [Background] Peralta I, Spooner DM. Genetic Improvement of Solanaceous Crops Volume 2: Tomato. CRC Press; 2006. https://books.google.com/books?hl=en&lr=&id=1m7RBQAAQBAJ&pgis=1. Accessed December 18, 2015
- [Background] Manach C., Brennan L, Drasgted L.O. Metabolomics to evaluate food intake and utilization in nutritional epidemiology. In: Metabolomics as a Tool in Nutritional Research, Woodhead publishing 2015. pp.167-196
- [Background] Kesse-Guyot E, Castetbon K, Touvier M, Hercberg S, Galan P. Relative validity and reproducibility of a food frequency questionnaire designed for French adults. Ann Nutr Metab. 2010;57(3-4):153-62. doi: 10.1159/000321680. Epub 2010 Nov 16. PMID 21079389
- [Derived] Vazquez-Manjarrez N, Weinert CH, Ulaszewska MM, Mack CI, Micheau P, Petera M, Durand S, Pujos-Guillot E, Egert B, Mattivi F, Bub A, Dragsted LO, Kulling SE, Manach C. Discovery and Validation of Banana Intake Biomarkers Using Untargeted Metabolomics in Human Intervention and Cross-sectional Studies. J Nutr. 2019 Oct 1;149(10):1701-1713. doi: 10.1093/jn/nxz125. PMID 31240312

DOCUMENTS (2):
  • Study Protocol (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03581955/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/55/NCT03581955/SAP_001.pdf